CLINICAL TRIAL: NCT04421066
Title: Histological, Genetic and Epigenetic Analysis of Procedures Related with Dental Implants
Status: Completed | Type: Observational
Sponsor: Simón Pardiñas López (Other)
Collaborators: NYU Langone Health (Other); Göteborg University (Other); University Hospital A Coruña (Other); Instituto de Investigacion Biomedica de A Coruna (Other)
Responsible Party: Sponsor-Investigator, Simón Pardiñas López, Director, Fundacion Clinica Pardinas
Organization: Fundacion Clinica Pardinas (Other)
Other Study IDs: 18-101718
Record Dates: First submitted 2020-06-01; First posted 2020-06-09 (Actual); Last update posted 2025-02-26 (Actual); Status verified 2025-02

CONDITIONS: Peri-Implantitis; Peri-implant Mucositis; Implant Complication; Implant Tissue Failure
MeSH Terms: conditions — Peri-Implantitis | interventions — Chewing Gum

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Biospecimen Retention: Samples With DNA — Gingival and bone samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Peri-implantitis: Patients with at least one dental implant diagnosed with peri-implantitis undergoing treatment for peri-implantitis as their standard of care will be included in this study.
  Interventions: Procedure: Gingival and bone sample collection
- Healthy: Patients with general good health and health gingiva undergoing extraction of wisdom tooth will be included in this study group.
  Interventions: Procedure: Healthy individuals

INTERVENTIONS:
Procedure: Gingival and bone sample collection — Gingival and bone samples will be collected from the sites affected by peri-implantitis during their surgical treatment of peri-implantitis or histological and epigenetic analysis.
  Groups: Peri-implantitis
Procedure: Healthy individuals — Gingival and bone samples will be collected from the extraction sites for histological and epigenetic analysis.
  Groups: Healthy

SUMMARY:
In this study genomic, proteomic and histological technologies for the search and characterization of epigenetic modifications and molecular or protein markers, useful in the diagnosis and progression of peri-implant diseases and prevention of implant failure will be used.

DETAILED DESCRIPTION:
Samples stored at the Biomedical Research Institute of A Coruña, Xerencia Integrated Management of A Coruña (University Hospital Center of A Coruña), belonging to the collection of the line of research "Oral Health and Systemic Relationship" with registration nº 2017/104 will be used for the realization of the present study.

Nucleic acid extraction and histological analysis of the samples will be performed to evaluate the functional epigenetic modifications associated with peri-implant diseases, in an exploratory manner.

ELIGIBILITY:
Inclusion Criteria:

* The subjects must have read, understood and signed an informed consent regarding the obtaining of biological samples and participation in the research line of "Oral Health and Systemic Relationship" existing in the Pardiñas Dental Medical Clinic and approved by the ethical committee.
* The subjects must be between 20-90 years of age.
* Subjects must be non-smokers or former smokers who have quit smoking for at least one year prior to enrollment in the study.

In addition to the general criteria listed, samples of a healthy periodontal subject must meet the following criteria when reviewing their medical and dental history :

-Subjects do not have or have had a history of periodontal disease, as described in the " 2017 World Workshop on the Classification of Periodontal and Peri- Implant Diseases and Conditions "

Samples from a subject with peri-implant disease must meet the following criteria:

-Samples of subjects who have at least one implant - supported prosthesis for at least 12 months and affected by peri- implant disease according to the " 2017 World Workshop on the Classification of Periodontal and Peri-Implant Diseases and Conditions "

Exclusion Criteria:

* Samples of pregnant or lactating women at the time of collection.
* Samples of subjects who were taking antibiotics within 1 month before collection of the sample.
* Samples of subjects with chronic use of non-steroidal anti-inflammatory drugs for more than 3 weeks at the time of sample collection. The use of aspirin in low doses (≤81 mg / day) will be allowed .
* Samples from subjects with disease in the mucosa in the area located around the site of sample collection.
* Samples of subjects with a systemic disease that would exclude the analysis (for example, severe medical problems, bone metabolism disorders, uncontrolled bleeding disorders, depressed immune system, diseases that require the periodic use of steroids, uncontrolled endocrine disorders) .
* Samples of subjects with a history of local irradiation therapy in the head / neck area.
* Samples of subjects with a history of having received treatment with intravenous or subcutaneous antiresorptive agents associated with osteonecrosis of the jaw, such as bisphosphonates.

Samples of subjects assigned to the healthy group that meet any of the following criteria will be excluded from participation in this study:

* Root fragments, pericoronaritis, endo-perio lesions, dental abscesses at the site of the biopsy.
* Presence of BOP in the sample collection site.

Peri- implant disease samples / Exclusion of Subjects

The samples of the subjects assigned to the peri- implant diseases group that meet any of the following criteria will be excluded from participation in this study if the implants were removed due to:

* Inadequate position of the implant.
* Subjects with implants previously treated surgically for peri- implant disease with antibiotics.

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: * Periodontally Healthy Subjects
  * Peri-implantitis Subjects
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2019-01-29 (Actual); Primary Completion 2021-10-21 (Actual); Study Completion 2022-06-20 (Actual)

PRIMARY OUTCOMES:
Differences in histological characteristics in peri-implantitis subjects compared to healthy subjects, ie, presence and amount of inflammatory cells and bacteria. | 1 day
  Gingival and blood samples collected from healthy subjects and subjects with peri-implantitis (including failing implants) will be used to determinate histological characteristics associated with peri-implantitis.
Differences in epigenetic characteristics analyzing DNA methylation in peri-implantitis subjects compared to healthy subjects. | 1 day
  Gingival and blood samples collected from healthy subjects and subjects with peri-implantitis (including failing implants) will be used to determinate epigenetic characteristics associated with peri-implantitis.

SECONDARY OUTCOMES:
Relation between peri-implant diseases and epigenetic modifications in terms of periodontal pocket depth. | 1 day
  To determine whether periodontal measurements PPD (in mm) are associated with epigenetic modifications.
Relation between peri-implant diseases and epigenetic modifications in terms of bleeding on probing. | 1 day
  To determine whether periodontal measurements bleeding on probing (BOP) (measured in percentage), are associated with epigenetic modifications.
Relation between peri-implant diseases and epigenetic modifications in terms of clinical attachment level. | 1 day
  To determine whether periodontal measurements CAL (clinical insertion level in mm), are associated with epigenetic modifications.
Relation between peri-implant diseases and epigenetic modifications in terms of plaque index. | 1 day
  To determine whether periodontal measurements plaque index (Sillness & Loe index)
Patient-reported outcome measures. | 1 day
  To determine whether patient-reported outcome measures (PROMs) are related to histological and epigenetic outcomes.
  Oral Health Impact Profile-14 (OHIP-14) assessed at study visit.

CONTACTS AND LOCATIONS:
Overall Officials: Simón Pardiñas López, DDS, MS, Principal Investigator — Fundación Clínica Pardiñas
Locations (1):
- Fundacion Clinica Pardiñas, A Coruña, Galicia, Spain

IPD SHARING:
Plan to Share IPD: Undecided